CLINICAL TRIAL: NCT05990491
Title: Pituitary Function After Recovery From Septic Shock Among ICU Survivors: A Prospective, Observational Study
Brief Title: Pituitary Function After Recovery From Septic Shock Among ICU Survivors
Status: Recruiting | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: A-05-PGI/IMP/87/2023
Record Dates: First submitted 2023-07-30; First posted 2023-08-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Shock, Septic; Pituitary Dysfunction; Hypopituitarism
Keywords: Septic shock; Post intensive care syndrome; Hypopituitarism
MeSH Terms: conditions — Shock, Septic; Hypopituitarism; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (8-10 ml) collected at the time of recruitment and at 6 months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic shock group: Patients 18-80 years of age who meet the definition of septic shock. Vasopressor requirement should be maintained for a period >24 hours and should require ICU stay for a duration of > 7 days. Patient should recover from shock and be planned for discharge from the ICU.
- Non-septic shock group: Patients 18-80 years of age who planned for discharge from the ICU.with stay for a duration of >7 days. Also, they should not have received vasopressor for.a period of >24 hours

SUMMARY:
Prolonged circulatory shock is associated with marked disturbances in vascular supply to the brain, and endothelial dysfunction which can lead to disseminated intravascular coagulation and microvascular thrombosis. Pituitary dysfunction is documented following post-partum hemorrhage, traumatic brain injury and subarachnoid hemorrhage, which also affect blood flow to the pituitary. However, there are no studies assessing pituitary function in the aftermath of recovery from shock. This will be a prospective observational study of patients admitted in Critical Care Medicine (CCM) ICU who have recovered from prolonged septic shock (Lasting for a period of > 24 hours). Blood samples of the participants will be estimated at the time of discharge from the ICU and at 6 months post discharge. Investigators will estimate fasting serum cortisol, TSH, Free T4, Testosterone (in males), Oestrogen (in females), LH, FSH, Prolactin, IGF-1 and plasma ACTH in all participants at both time points (at the time of ICU discharge and at 6-months follow-up). Participants who have borderline serum cortisol values (138-400 nmol/l) will be subjected to 250ug ACTH stimulation test. Expected outcome of the proposed study is to know proportion of patients having pituitary hormone axis dysfunction. Investigators will also look for pituitary dysfunction persist or revert, or there are new onset dysfunction at 6 month follow up. This would have major implications in the follow up and management of ICU survivors.

DETAILED DESCRIPTION:
The pituitary gland receives its arterial blood supply from the superior and inferior hypophyseal arteries, which arise from the internal carotid artery. The infundibulum, the median eminence and the pars tuberalis are supplied by the superior hypophyseal artery and the posterior lobe by the inferior hypophyseal artery. By contrast, the pars distalis (anterior pituitary) is mainly supplied by the venous system. The long portal system, arising from the capillary plexus around the median eminence, and the short portal system arising from the posterior pituitary account for 70% and 30% respectively, of the total blood supply to the anterior pituitary gland. This unique circulation allows the pars distalis to receive humoral signals from the hypothalamus and the posterior pituitary; however, it renders the pituitary susceptible to ischemia due to hypotension, hypovolemia and vascular thrombosis.

The prototype illness where pituitary necrosis leads to pituitary dysfunction is post-partum pituitary necrosis (Sheehan syndrome). The pituitary gland becomes vulnerable to changes in blood flow during and shortly after pregnancy owing to the increased size of the gland, leading to both increased demand and compression of the vasculature of the gland. In addition, pregnancy is a thrombophilic state which increases risk for intravascular thrombosis. Hypotension secondary to post-partum hemorrhage causes pituitary necrosis and leads to hypopituitarism. Vascular insults to the pituitary are also implicated in other forms of pituitary damage, such as following traumatic brain injury, following snakebite envenomation, subarachnoid hemorrhage and hemorrhagic shock.

Circulatory shock replicates many of the pathophysiological processes described above. Clinical classifications of shock include hypovolemic, cardiogenic, distributive (septic), and obstructive types. While the pathophysiology of each type of shock is different and complex, the final common pathway is poor perfusion, anaerobic metabolism, lactic acidosis, and release of inflammatory mediators with resultant tissue damage. Sepsis and septic shock are often complicated by Disseminated Intravascular Coagulation (DIC) which leads to widespread microvascular thrombosis. Hypotension leads to reduced blood flow to the hypothalamo-pituitary unit and all these factors may lead on to ischemia and infarction of the hypothalamo-pituitary unit. Patients who recovered post cardiac arrest suffer an extreme form of this insult where blood flow to the brain is almost entirely cut off for a period of time, followed by reperfusion.

Post ICU Care Syndrome (PICS) is estimated to occur in 30-80% of patients post discharge from the intensive care unit. Many of the manifestations of Post ICU Care Syndrome (PICS), such as fatigue, cognitive dysfunction, neuromuscular weakness, amenorrhea and sexual dysfunction overlap with those seen in hypopituitarism. However, there is no literature describing the role of pituitary dysfunction in these patients.

Based on the above evidence, we hypothesize that patients who recover from severe shock may have hypothalamic-pituitary damage leading to hypopituitarism. Due to the current lack of literature on this topic, we propose to study pituitary function in ICU survivors who recovered from the septic shock.

The primary objective is to study the prevalence of dysfunction of various pituitary hormone axes at the time of ICU discharge in participants who recovered from the septic shock. The secondary objective is to look for the recovery of pituitary function or new onset pituitary dysfunction at 6 months post-discharge from the ICU, in these included participants.

This will be a prospective, observational study of participants undergoing treatment for septic shock in the Department of Critical Care Medicine (CCM), SGPGIMS, Lucknow.

Details of premorbid conditions, precipitating illness, clinical parameters and treatments provided to the participants will be recorded. Levels of pituitary hormones [Cortisol (Basal and stimulated), ACTH, IGF-1, LH, FSH, Testosterone (in males), Estradiol (in females), Prolactin, TSH and free T4] will be assessed in fasting state, prior to discharge from the ICU. Participants will be interviewed telephonically at 3 months post-discharge to assess quality of life using the SF-36 questionnaire and for symptoms suggestive of hypopituitarism. At 6 months post-discharge, the various pituitary hormone levels [Cortisol (Basal and stimulated), ACTH, IGF-1, LH, FSH, Testosterone (in males), Estradiol (in females), Prolactin, TSH and free T4] will be assessed again along with assessment of quality of life using SF-36. Any pituitary hormone deficiency identified on testing will be evaluated and managed as per standard practice.

Investigators aim to include 90 participants in the study. Continuous variables will be presented in mean and standard deviation (SD) or median (interquartile range) depending upon normality status. Independent samples t test (for independent groups) / Paired t test (paired groups) or their non-parametric counterparts will be used to compare the means or medians between the groups, respectively. Categorical variables will be presented in number (%) and will be compared by Chi square test / Fisher exact test, as appropriate. One-way Repeated Measures ANOVA or Friedman test will be used to compare the means or medians over the time as appropriate. Binary logistic regression analysis will be used to assess the factors associated with pituitary dysfunction among the study participants.

ELIGIBILITY:
Inclusion Criteria:

Septic shock group:

* Patients 18-80 years of age who meet the definition of septic shock.
* Vasopressor requirement should be maintained for a period > 24 hours and should require ICU stay for a duration of > 7 days.
* Patient should recover from shock and be planned for discharge from the ICU

Non-septic shock group

* Patients 18-80 years of age who planned for discharge from the ICU.with stay for a duration of >7 days.
* Also, they should not have received vasopressor for.a period of >24 hours

Exclusion Criteria:

* Patients who refuse to provide consent.
* Age <18 years or > 80 years of age.
* Pregnancy or immediate post-partum (< 6 months post-delivery).
* Chronic kidney disease (Stage 5), chronic liver disease (CHILD B or C), severe Chronic obstructive pulmonary disease, Chronic heart failure.
* Patients with pre-existing hypopituitarism on replacement.
* Past history of severe post-partum hemorrhage requiring blood transfusion, traumatic brain injury, subarachnoid hemorrhage, pituitary tumor/surgery, snake bite envenomation and meningo-encephalitis.
* Patients who have been on > 5 mg prednisolone equivalent for a period of more than 2 weeks at any time in the previous 6 months before admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to critical care medicine intensive care unit at Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow who meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pituitary dysfunction at discharge | Immediately before the ICU discharge
  Frequency of dysfunction of various hypothalamo-pituitary hormone axes

SECONDARY OUTCOMES:
Pituitary dysfunction at 6 months | Six months after the ICU discharge
  Frequency of dysfunction of various hypothalamo-pituitary hormone axes on follow up

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Yadav, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences; Mohan Gurjar, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences; Jayakrishnan C, DM, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences
Locations (2):
- India (2):
  - Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh
  - Department of Endocrinology, SGPGIMS, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No